CLINICAL TRIAL: NCT01726231
Title: Evaluation of Abdominal Wall Lifting During Laparoscopic Direct Trocar Insertion
Status: Completed | Type: Observational
Sponsor: Bagcilar Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: BEH GynObs-2
Record Dates: First submitted 2012-11-09; First posted 2012-11-14 (Estimated); Last update posted 2013-12-25 (Estimated); Status verified 2013-12

CONDITIONS: Other Surgical Procedures
Keywords: Laparoscopic access; Abdominal wall lifting; Direct trocar insertion; Safety endoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
In laparoscopy, over %50 of the all complications occur during establishment of the pneumoperitoneum. Lifting of the anterior abdominal wall is aimed to increase the distance between the abdominal wall and the intrabdominal structures. Elevation of the anterior abdominal wall is recommended for the access to peritoneal cavity in literatures however the benefit exactly has not proved. This study aimed to determine the distance from anterior abdominal wall to intraperitoneal structures during lifting of the abdominal wall, to represent this distance -on the average- generate the safe range whether or not and compare with this distance and patient's age, BMI and parity.

DETAILED DESCRIPTION:
40 patients who undergoing laparoscopic surgery for various indications are enrolled in the study. The telescope is inserted at second trocar place and the distances between anterior abdominal wall and visceral organs are measured with plastic hysterometry during maximal elevation of the abdominal wall.

ELIGIBILITY:
Inclusion Criteria:

* the patients who performed laparoscopic surgery

Exclusion Criteria:

* the patients who suspected pregnancy
* large scale intrabdominal mass

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: the patiens undergoing laparoscopic surgery for various indications
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2012-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure of this study is to determine the distance in centimeters from anterior abdominal wall to intraperitoneal visceral structures during lifting of the abdominal wall with plastic hysterometry. | 2-3 months

CONTACTS AND LOCATIONS:
Overall Officials: TANER A USTA, M.D., Principal Investigator — Bagcilar Training and Research Hospital, Istanbul, Turkey
Locations (1):
- Bagcilar Training and Research Hospital, Istanbul, Turkey (Türkiye)